CLINICAL TRIAL: NCT00429442
Title: A Double Blind, Randomised, Placebo Controlled Study Investigating Simvastatin as an add-on Treatment to Copaxone for the Treatment of Relapsing Multiple Sclerosis in Patients Treated With Copaxone for at Least 3 Months
Brief Title: Simvastatin as an add-on Treatment to Copaxone for the Treatment of Relapsing Multiple Sclerosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Anna Tsakiri (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Anna Tsakiri, MD, PhD, Glostrup University Hospital, Copenhagen
Organization: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CoSim-01; EudraCT number 2006-001827-21
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Simvastatin; CNS Inflammation; Copaxone
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Simvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Simvastatin — 80 mg once daily
  Arms: 1
Drug: placebo — calcium tablets once daily
  Arms: 2

SUMMARY:
A Double Blind, Randomised, Placebo Controlled Study Investigating Simvastatin as an add-on Treatment to Copaxone for the Treatment of Relapsing Multiple Sclerosis in patients treated with Copaxone for at least 3 months

DETAILED DESCRIPTION:
This is a double blind, placebo controlled, randomised, phase 3 study. Patients that have been treated with Copaxone for at least 6 months at the screening visit will be randomised for treatment with simvastatin or placebo as an add-on to their Copaxone treatment. Patients will start treatment with 40 mg peroral simvastatin daily (or an apparently identical placebo) for one month. Hereafter, patients will escalate dosage to 80 mg daily. The patients will be examined clinically at screening, baseline and at 3, 6 and 12 months. Blood samples for immunology will be performed at baseline and at 1, 3, 6 and 12 months. Blood samples for safety assessments will be performed at all study visits. MRI will be performed (T1-weighted and T2-weighted) at baseline and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* A patient may be included if s/he fulfils all criteria mentioned below:

  * The patient must give written informed consent prior to any study related activities. Study related activities are any procedures that would not have been performed during normal management of the patient.
  * Is between the age of 18 and 60 years (both included).
  * Suffers from definite relapsing-remitting MS according to Poser criteria (CDMS or LSDMS) 21 or definite MS according to McDonald criteria 22.
  * Has a disability equivalent to an EDSS of 6.5 or less 20.
  * Has shown clinical activity defined as at least one reported or documented relapse within the last year or two reported or documented relapses within the last two years.
  * Has been treated with Copaxone for at least 3 months.
  * The patient must be prepared to and considered able to follow the protocol during the whole study period and to attend the planned visits, even if the treatment has to be withdrawn.

Exclusion Criteria:

* The patient must not be included if any of the criteria mentioned below are fulfilled:

  * Any condition that might give rise to similar symptoms as MS.
  * Has received treatment with glucocorticoids or ACTH later than one month prior to inclusion into the study, i.e. at the screening visit.
  * Has experienced the onset of a relapse within one month prior to inclusion into the study, i.e. at the screening visit.
  * Has suffered from major depression.
  * Has received immuno-suppressive treatment in the 6 months prior to screening.
  * Alcohol or drug dependency.
  * Has cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV).
  * Significant hypertension (BP > 180/110 mmHg).
  * Has renal insufficiency defined as serum creatinine > 1.5 times the upper normal reference limit.
  * ASAT and/or ALAT more than 1.5 times the normal upper reference limit.
  * Leucopaenia < 2.5 x 109/L or thrombopaenia < 100 x109/L.
  * Any medical illness requiring treatment with systemic corticosteroids.
  * Any systemic disease that can influence the patient's safety and compliance, or the evaluation of the disability.
  * Women who are pregnant, breast-feeding or have the possibility for pregnancy during the study. To avoid pregnancy, women have to be postmenopausal, surgically sterile, sexually inactive or practice reliable contraception (contraceptive pill, intrauterine device, administration of deposit of progestins, subcutaneous implants, contraception ring, transdermal deposit plaster).
  * Known or suspected allergy to study product or related products.
  * Participation in any other studies, involving other investigational product, within 30 days prior to participating in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Number of new and/or enlarging lesions on T2- weighted MRI based on MRI done 12 months following baseline compared with MRI done at baseline. | one year

SECONDARY OUTCOMES:
Changes in the EDSS score between baseline and 12 months after baseline. | one year
Changes in the MFSC score between baseline and 12 months after baseline. | one year
Number of documented relapses after baseline. | one year
Changes in immunological parameters | one year
Regulation of immunological activation. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jette L Frederiksen, DMSC, Principal Investigator — Department of Neurology, Glostrup Hospital, Denmark
Locations (1):
- Department of Neurology, Glostrup University Hospital, Glostrup Municipality, Glostrup, Denmark